CLINICAL TRIAL: NCT00213109
Title: Open Trial of Miglitol in Type 1 Diabetic Patients With Insulin Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG1006
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: alpha-glucosidase inhibitor,Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — miglitol

INTERVENTIONS:
Drug: Miglitol

SUMMARY:
The purpose of this study is evaluate the clinical efficacy and safety of Miglitol in patients with Type1 Diabetes Mellitus treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type1 Diabetes
* Criteria of postprandial glucose and HbA1c are met

Exclusion Criteria:

* Type2 Diabetes
* Patients with antidiabetic drugs
* The other exclusion criteria are met

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Promotion Group, Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (7):
- Japan (7):
  - Chiba
  - Fukuoka
  - Gifu
  - Ibaraki
  - Kanagawa
  - Kumamoto
  - Ōita